CLINICAL TRIAL: NCT06178627
Title: A Multi-center, Prospective, Randomized Trial of Amphotericin B in the Initial Antifungal Therapy for Non-HIV Cryptococcal Meningitis Patients
Brief Title: Amphotericin B for Non-HIV Cryptococcal Meningitis Patients
Acronym: ABNCM
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Li-Ping Zhu, Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Huashan Hospital ID
Record Dates: First submitted 2023-12-04; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Cryptococcal Meningitis; Antifungal Agents
Keywords: Cryptococcal Meningitis; Antifungal agents; amphotericin B; non-HIV
MeSH Terms: conditions — Meningitis, Cryptococcal | interventions — Amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal dose amphotericin B (0.7 mg/kg/d) (Active Comparator): Study regimen 1: amphotericin B 0.7 mg/kg/day i.v. plus flucytosine for 4 weeks
  Interventions: Drug: Amphotericin B 0.7 mg/kg/day i.v. combined with flucytosine four times per day orally for the first 4 weeks.
- Low dose amphotericin B (0.5 mg/kg/d) (Experimental): Amphotericin B 0.5 mg/kg/day i.v. plus flucytosine for 4 weeks
  Interventions: Drug: Amphotericin B 0.5 mg/kg/day i.v. combined with flucytosine four times per day orally for the first 4 weeks.

INTERVENTIONS:
Drug: Amphotericin B 0.5 mg/kg/day i.v. combined with flucytosine four times per day orally for the first 4 weeks. — Different amphotericin B dosage
  Arms: Low dose amphotericin B (0.5 mg/kg/d)
Drug: Amphotericin B 0.7 mg/kg/day i.v. combined with flucytosine four times per day orally for the first 4 weeks. — Different amphotericin B dosage
  Arms: Normal dose amphotericin B (0.7 mg/kg/d)

SUMMARY:
Cryptococcus neoformans and C. gatti are important causes of central nervous system (CNS) infections with significant mortality, remaining a great public health challenge worldwide. Commonly seen as an opportunistic infection in adults with HIV/AIDS, cryptococcal meningitis (CM) accounts for 15% of HIV-related mortality globally [1]. In addition, a growing number of non-HIV CM patients have been observed in recent years with fatality approaching 30% in some areas [2,3]. It occurs in both those with natural or iatrogenic immunosuppression, as well as the apparently immunocompetent individuals. Approximately 65-70% of non-HIV CM patients were without any predisposing factors, particularly in the East Asia [4,5]. With the increasing number of hematopoietic stem cell transplantation, solid organ transplantation recipients and administration of immunosuppressive and corticosteroids agents, this illness will assume even greater public health significance.

Current Infectious Disease Society of America (IDSA) guideline suggest the use of combination antifungal therapy: normal dose amphotericin (0.7-1mg/kg/day) combined with flucytosine for a minimum of 4 weeks, followed by fluconazole (600-800 mg/day) for a minimum of 10 weeks in total for HIV patients [6]. However, for non-HIV and immunocompetent patients, the treatment remains controversial. IDSA guideline recommended that the treatment of non-HIV patients could refer to the treatment of HIV patients. That is, amphotericin B combined with flucytosine is still administered in the induction period. However, as amphotericin B have nonspecific effect on ergosterol, it has strong side effects (hepatorenal toxicity, electrolyte disorder, anemia, ventricular fibrillation, etc.). Therefore, the dose of amphotericin B may not be appropriate for Asian patients due to the different drug metabolism and pharmacokinetic. In the prospective studies of Bennett[7] and Dismuke[8], low dose amphotericin B (0.3 mg/kg/d) combined with flucytosine achieved response rates of 66% and 85% at 6 weeks, respectively. A similar conclusion was also extracted from a large multicenter retrospective study that low dose amphotericin B (<0.7 mg/kg/d) combined with flucytosine for a minimum of 2 weeks, followed by fluconazole could achieve a response rate of 84%, indicating that the efficacy of low dose amphotericin B (< 0.7 mg/kg/d) may be equivalent with normal dose in non-HIV patients. Therefore, we plan to conduct a prospective, multicenter, open-label randomized controlled study to compare the efficacy and safety of normal dose amphotericin B (0.7 mg/kg/ d) and low dose amphotericin B (0.5 mg/kg/d) in the initial antifungal treatment for non-HIV cryptococcal meningitis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years
2. HIV antibody negative
3. Cryptococcal meningitis defined as a syndrome consistent with CM and one or more of: 1) positive CSF India ink (budding encapsulated yeasts), 2) C.neoformans cultured from CSF or blood, 3) positive cryptococcal antigen Lateral Flow Antigen Test (LFA) in CSF, 4) positive brain tissue representing Cryptococcus
4. Having no severe immunocompromised conditions
5. Informed consent to participate given by patient or acceptable representative

Exclusion Criteria:

1. Previously cryptococcal disease
2. Currently receiving treatment for cryptococcal meningitis and having received ≥72 hours of anti-cryptococcal meningitis therapy in 96 hours
3. Creatinine clearance lower than 80 ml/min
4. Liver dysfunction (defined as ALT or AST > 2×ULN and bilirubin > 1.5×ULN, or ALT or AST > 3×ULN, or bilirubin > 2×ULN)
5. Liver cirrhosis or chronic liver failure
6. Pregnancy or breast-feeding
7. Known allergy to study drugs
8. Failure to consent - the patient, or if they are incapacitated, their responsible relative, declines to enter the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-08-13 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Mortality rate at 4 weeks after randomization. | 4 weeks
  The primary end point was mortality rate at 4 weeks after randomization. Mortality was treated as a binary variable, and the generalized linear model (GLM) was used for non-inferiority test. Point estimation and one-sided 95% confidence interval (CI) estimation of mortality difference between the two groups will be performed. If the upper limit value of 95% CI is less than 0.10 of the non-inferiority margin, the research result is considered to be in line with the non-inferiority margin. Kaplan-meier was used to draw the four week survival curves of the two groups, and log rank method was used to test the survival curves. Cox proportional hazard regression model was used to analyze the risk of death (HR) and 95% CI of the two groups. Sensitivity analysis: in the above analysis, the patients who lost the follow-up within 4 weeks were excluded for sensitivity analysis; The above non inferiority test GLM analysis and cox model included confounding variables (baseline Log10 fungal load, w

SECONDARY OUTCOMES:
EFA rate at 2 weeks after randomization | 2 weeks
  All recorded longitudinal quantitative fungal count measurements up to day 35 (allowing for some delays in the day 28 measurements) will be included in the analysis. EFA will be modeled based on a linear mixed effects model with longitudinal log10-CSF quantitative culture fungal counts as the outcome, interaction terms between the treatment groups and the time since enrolment of the measurement as fixed covariates and random patient-specific intercepts and slopes. The lowest measurable quantitative count is 5 CFU/ml and values below the detection limit (which correspond to recorded values of 0) will be treated as <4.5 CFU/ml, i.e. non-detectable measurements will be treated as left-censored longitudinal observations in the analysis. Based on this model, EFA will be compared between the 3 treatment arms in all patients (intention to treat), in the per-protocol population, and subgroups defined by immune status (immunocompromised; immunocompetent) and baseline fungal burden.
urvival until 2 weeks, 10 weeks and 6 months after randomization | up to 6 months
  Overall survival will be visualized using Kaplan-Meier curves and modeled using the Cox proportional hazards regression model with stratification by immune status. In addition, survival will be modeled with a multivariable Cox regression model including the following covariates in addition to the treatment group: baseline log10-fungal load, Glasgow coma score less than 15 (yes or no) and immune status.
Disability at 10 weeks and 6 months | up to 6 months
  The disability score at week 10 follow-up is defined as the higher (worse) of " the three simple questions" and the modified Rankin score assessed at that time point, and will be categorized as good outcome, intermediate disability, severe disability, or death (in case the patient died before 10 weeks) as previously described (wellcome-45). The ordinal 10-week score ("good">"intermediate">"severe"> "death") will be compared between the 3 arms with a proportional odds logistic regression model depending on the treatment arm. The result will be summarized as a cumulative odds ratio with corresponding 95% confidence interval and P value. Patients lost to follow up will be analyzed according to their last recorded disability status. If the rate of patients lost to follow-up exceeds 10%, we will also perform an alternative analysis based on multiple imputation of missing values. The three simple questions and the modified Rankin score are listed in Appendix 4.
Adverse events | 4 weeks
  The frequency of serious and grade 3&4 adverse reactions as well as the frequency of specific adverse events will be summarized (both in terms of the total number of events as well as the number of patients with at least one event). The proportion of patients with at least one such event (overall and for each specific event separately) will be summarized and (informally) compared between the 3 treatment groups based on χ2 test or Fisher's exact test, as appropriate. 6) Visual deficit at 10 weeks and 6 months
Visual deficit at 10 weeks and 6 months | up to 6 months
  The visual acuity at 10 weeks is recorded on a 6 point scale (see Appendix 5) and will be summarized by treatment arm for each eye separately, and overall where "overall" is defined as the worst recorded acuity of either eye. The odds of having "normal acuity" (amongst all surviving patients with a visual assessment) will be informally compared between the treatment arms with a logistic regression model adjusted for immune status.
Time to new neurological event or death until 10 weeks | up to 10 weeks
  The time to the first new neurological event or death until 10 weeks will be analyzed in the same way as overall survival. Longitudinal measurements of intracranial pressure during the first 2 weeks will be modeled using a mixed effect model as described for the primary outcome.
Rate of IRIS at 10 weeks and 6 months | up to 6 months
  The rate of IRIS and the rate of relapse (defined as antifungal treatment intensification or re-treatment) will be modeled with cause-specific proportional hazards models with treatment as the only covariate and stratification by immune status.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - The Fourth People's Hospital of Nanning, Nanning

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lortholary O, Dromer F, Mathoulin-Pelissier S, Fitting C, Improvisi L, Cavaillon JM, Dupont B; French Cryptococcosis Study Group. Immune mediators in cerebrospinal fluid during cryptococcosis are influenced by meningeal involvement and human immunodeficiency virus serostatus. J Infect Dis. 2001 Jan 15;183(2):294-302. doi: 10.1086/317937. Epub 2000 Dec 8. PMID 11110651
- [Background] Jiang YK, Wu JQ, Zhao HZ, Wang X, Wang RY, Zhou LH, Yip CW, Huang LP, Cheng JH, Chen YH, Li H, Zhu LP, Weng XH. Genetic influence of Toll-like receptors on non-HIV cryptococcal meningitis: An observational cohort study. EBioMedicine. 2018 Nov;37:401-409. doi: 10.1016/j.ebiom.2018.10.045. Epub 2018 Oct 23. PMID 30366814
- [Background] Haddow LJ, Colebunders R, Meintjes G, Lawn SD, Elliott JH, Manabe YC, Bohjanen PR, Sungkanuparph S, Easterbrook PJ, French MA, Boulware DR; International Network for the Study of HIV-associated IRIS (INSHI). Cryptococcal immune reconstitution inflammatory syndrome in HIV-1-infected individuals: proposed clinical case definitions. Lancet Infect Dis. 2010 Nov;10(11):791-802. doi: 10.1016/S1473-3099(10)70170-5. PMID 21029993
- [Background] Chau TT, Mai NH, Phu NH, Nghia HD, Chuong LV, Sinh DX, Duong VA, Diep PT, Campbell JI, Baker S, Hien TT, Lalloo DG, Farrar JJ, Day JN. A prospective descriptive study of cryptococcal meningitis in HIV uninfected patients in Vietnam - high prevalence of Cryptococcus neoformans var grubii in the absence of underlying disease. BMC Infect Dis. 2010 Jul 9;10:199. doi: 10.1186/1471-2334-10-199. PMID 20618932
- [Background] Thwaites GE, Nguyen DB, Nguyen HD, Hoang TQ, Do TT, Nguyen TC, Nguyen QH, Nguyen TT, Nguyen NH, Nguyen TN, Nguyen NL, Nguyen HD, Vu NT, Cao HH, Tran TH, Pham PM, Nguyen TD, Stepniewska K, White NJ, Tran TH, Farrar JJ. Dexamethasone for the treatment of tuberculous meningitis in adolescents and adults. N Engl J Med. 2004 Oct 21;351(17):1741-51. doi: 10.1056/NEJMoa040573. PMID 15496623
- [Background] Beardsley J, Wolbers M, Kibengo FM, Ggayi AB, Kamali A, Cuc NT, Binh TQ, Chau NV, Farrar J, Merson L, Phuong L, Thwaites G, Van Kinh N, Thuy PT, Chierakul W, Siriboon S, Thiansukhon E, Onsanit S, Supphamongkholchaikul W, Chan AK, Heyderman R, Mwinjiwa E, van Oosterhout JJ, Imran D, Basri H, Mayxay M, Dance D, Phimmasone P, Rattanavong S, Lalloo DG, Day JN; CryptoDex Investigators. Adjunctive Dexamethasone in HIV-Associated Cryptococcal Meningitis. N Engl J Med. 2016 Feb 11;374(6):542-54. doi: 10.1056/NEJMoa1509024. PMID 26863355
- [Background] Day JN, Chau TTH, Wolbers M, Mai PP, Dung NT, Mai NH, Phu NH, Nghia HD, Phong ND, Thai CQ, Thai LH, Chuong LV, Sinh DX, Duong VA, Hoang TN, Diep PT, Campbell JI, Sieu TPM, Baker SG, Chau NVV, Hien TT, Lalloo DG, Farrar JJ. Combination antifungal therapy for cryptococcal meningitis. N Engl J Med. 2013 Apr 4;368(14):1291-1302. doi: 10.1056/NEJMoa1110404. PMID 23550668
- [Background] Zhao HZ, Wang RY, Wang X, Jiang YK, Zhou LH, Cheng JH, Huang LP, Harrison TS, Zhu LP. High dose fluconazole in salvage therapy for HIV-uninfected cryptococcal meningitis. BMC Infect Dis. 2018 Dec 12;18(1):643. doi: 10.1186/s12879-018-3460-7. PMID 30541454
- [Background] Perfect JR, Dismukes WE, Dromer F, Goldman DL, Graybill JR, Hamill RJ, Harrison TS, Larsen RA, Lortholary O, Nguyen MH, Pappas PG, Powderly WG, Singh N, Sobel JD, Sorrell TC. Clinical practice guidelines for the management of cryptococcal disease: 2010 update by the infectious diseases society of america. Clin Infect Dis. 2010 Feb 1;50(3):291-322. doi: 10.1086/649858. PMID 20047480
- [Background] Chen J, Varma A, Diaz MR, Litvintseva AP, Wollenberg KK, Kwon-Chung KJ. Cryptococcus neoformans strains and infection in apparently immunocompetent patients, China. Emerg Infect Dis. 2008 May;14(5):755-62. doi: 10.3201/eid1405.071312. PMID 18439357
- [Background] Zhu LP, Wu JQ, Xu B, Ou XT, Zhang QQ, Weng XH. Cryptococcal meningitis in non-HIV-infected patients in a Chinese tertiary care hospital, 1997-2007. Med Mycol. 2010 Jun;48(4):570-9. doi: 10.3109/13693780903437876. PMID 20392150
- [Background] Brizendine KD, Baddley JW, Pappas PG. Predictors of mortality and differences in clinical features among patients with Cryptococcosis according to immune status. PLoS One. 2013;8(3):e60431. doi: 10.1371/journal.pone.0060431. Epub 2013 Mar 26. PMID 23555970
- [Background] Rajasingham R, Smith RM, Park BJ, Jarvis JN, Govender NP, Chiller TM, Denning DW, Loyse A, Boulware DR. Global burden of disease of HIV-associated cryptococcal meningitis: an updated analysis. Lancet Infect Dis. 2017 Aug;17(8):873-881. doi: 10.1016/S1473-3099(17)30243-8. Epub 2017 May 5. PMID 28483415